CLINICAL TRIAL: NCT07016802
Title: A Randomized, Double-Blind, Placebo and Positive Drug-Controlled, Single-Dose, Dose-Escalation Phase I Clinical Study of GenSci134 Injection in Healthy Adults
Brief Title: A Clinical Study of GenSci134 in Healthy Male Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GenSci134-101
Record Dates: First submitted 2025-05-30; First posted 2025-06-12 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GenSci134 (Experimental)
  Interventions: Drug: GenSci134
- GenSc134 Placebo (Placebo Comparator)
  Interventions: Drug: GenSci134 Placebo
- Recombinant Human Growth Hormone Injection (Norditropin®) (Active Comparator)
  Interventions: Drug: Recombinant Human Growth Hormone Injection (Norditropin®)

INTERVENTIONS:
Drug: GenSci134 — only one dose of GenSci134 and GenSci134 Placebo to be given, subcutaneous , 7 dose levels will be assigned.
  Arms: GenSci134
Drug: GenSci134 Placebo — only one dose of GenSci134 and GenSci134 Placebo to be given, subcutaneous , 7 dose levels will be assigned.
  Arms: GenSc134 Placebo
Drug: Recombinant Human Growth Hormone Injection (Norditropin®) — A single dose of 0.2 mg/day, administered once daily (QD) for 28 consecutive days.
  Arms: Recombinant Human Growth Hormone Injection (Norditropin®)

SUMMARY:
To check how safe and well-tolerated a single subcutaneous injection of GenSc134 is in healthy male volunteers

DETAILED DESCRIPTION:
GenSci134 was tested in 7 predetermined dose groups with placebo and positive drug controls to explore the dosage, and to assess its safety, tolerability, pharmacokinetic (PK) characteristics, pharmacodynamic (PD) characteristics, immunogenicity, and exploratory endpoints in 64 healthy adult male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male subjects aged 18-45 years (inclusive of boundary values);
* Body Mass Index (BMI): 19.0-24.0 kg/m² (inclusive of boundary values);
* Good health status;
* Able to understand and willing to sign the Informed Consent Form (ICF), and comply with study requirements and restrictions.

Exclusion Criteria:

* Subjects with significant medical history or clinical manifestations determined by the investigator;
* History of hypersensitivity, intolerance, or allergy to any drug, compound, food, or other substances, or known allergy to any excipients of the study drug;
* History of neurological or psychiatric disorders, or subjects with impaired consciousness or cognitive dysfunction;
* Subjects with clinically significant abnormalities, including but not limited to vital signs or laboratory test results that are abnormal and clinically significant;
* Subjects with immunodeficiency or immunosuppressive diseases at screening;
* Subjects who have undergone major surgery within 12 months prior to screening;
* Subjects with a history of neoplastic diseases;
* Subjects who have participated in any other clinical trial of drugs or medical devices and have used the investigational medicinal product within 28 days or 5 half-lives (whichever is longer) before dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events | 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Dongyang LIU, PHD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China